CLINICAL TRIAL: NCT03701555
Title: A Phase 1, Four-Part Study to Assess the Safety, Tolerability, Pharmacokinetics, and Gluten Degradation Activity of PvP001, PvP002, and PvP003 in Healthy Adult Volunteers and to Assess the Safety, Tolerability, and Pharmacokinetics of PvP001 and PvP002 in Adults With Celiac Disease
Brief Title: A Study of PVP001, PVP002, and PVP003 in Healthy Adults and PVP001 and PVP002 in Adults With Celiac Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: PvP-102-01
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Results first posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2022-06

CONDITIONS: Digestive System Disease
MeSH Terms: conditions — Digestive System Diseases | interventions — Maximum Tolerated Dose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Part 1, Cohort 1A-1 to 1D-1 Healthy Participants (Experimental): A single dose of PvP001 placebo, PvP001 100 mg, PvP001 300 mg, or PvP001 900 mg will be administered in ascending order to healthy participants in Cohorts 1A-1, 1B-1, 1C-1, and 1D-1.
  Interventions: Other: PvP001 placebo; Drug: PvP001 100 mg; Drug: PvP001 300 mg; Drug: PvP001 900 mg
- Part 1, Cohort 1E-1 Healthy Participants (Experimental): A single dose of the maximum feasible dose (MFD) of PvP002 will then be administered to healthy participants in Cohort 1E-1.
  Interventions: Drug: Maximum Feasible Dose (MFD) of PvP002
- Part 1, Cohort 1A-2 - 1D-2 Celiac Disease (CeD) (Experimental): A single dose of PvP001 placebo, PvP001 100 mg, PvP001 300 mg, or PvP001 900 mg will be administered in ascending order to participants with CeD in Cohorts 1A-2, 1B-2, 1C-2, and 1D-2.
  Interventions: Other: PvP001 placebo; Drug: PvP001 100 mg; Drug: PvP001 300 mg; Drug: PvP001 900 mg
- Part 1, Cohort 1E-2 CeD (Experimental): A single dose of the MFD of PvP002 will then be administered to participants with CeD in Cohort 1E-2.
  Interventions: Drug: Maximum Feasible Dose (MFD) of PvP002
- Part 2, Cohort 2A - Cohort 2C Healthy Participants (Experimental): Participants will be blinded to the PvP001 dose (placebo or MTD of PvP001) and will also receive MTD of PvP001 following 7 days of PPI treatment.
  Interventions: Other: PvP001 placebo; Drug: Maximum Tolerated Dose (MTD) of PvP001; Drug: MTD of PvP001 following 7 days of PPI treatment
- Part 2, Cohort 2D Healthy Participants (Experimental): Participants will receive PvP001 placebo or MFD of PvP001.
  Interventions: Other: PvP001 placebo; Drug: Maximum Tolerated Dose (MTD) of PvP001
- Part 2, Cohort 2E Healthy Participants (Experimental): Participants will receive PvP002 placebo or MFD of PvP002.
  Interventions: Drug: Maximum Feasible Dose (MFD) of PvP002; Other: PvP002 placebo
- Part 2, Cohort 2F- Cohort 2H Healthy Participants (Experimental): Participants will receive the PvP001 placebo and either 300 mg or 600 mg of PvP001.
  Interventions: Other: PvP001 placebo; Drug: PvP001 300 mg; Drug: PvP001 600 mg
- Part 2, Cohort 2I and Cohort 2J Healthy Participants (Experimental): Participants will receive the PvP001 placebo and 900 mg of PvP001.
  Interventions: Other: PvP001 placebo; Drug: PvP001 900 mg
- Part 3, Cohorts 3A and 3B Healthy Participants (Experimental): Participants will receive single dose of PvP003 placebo and 600 mg of PvP003 with pretreatment buffer solution before a standardized 1 gm gluten-containing study meal.
  Interventions: Drug: PvP003 placebo; Drug: PvP003
- Part 3, Cohorts 3C and 3D Healthy Participants (Experimental): Participants will receive single dose of PvP003 placebo and 600 mg of PvP003 without pretreatment buffer solution before a standardized 1 gm gluten-containing study meal.
  Interventions: Drug: PvP003 placebo; Drug: PvP003
- Part 3, Cohorts 3E and 3F Healthy Participants (Experimental): Participants will receive single dose of PvP003 placebo and 600 mg of PvP003 without pretreatment buffer solution after an approximately 50 milliliter (mL) portion of a standardized 1 gm gluten-containing study meal.
  Interventions: Drug: PvP003 placebo; Drug: PvP003
- Part 3, Cohorts 3G and 3H Healthy Participants (Experimental): Participants will receive single dose of PvP003 placebo and 600 mg of PvP003 without pretreatment buffer solution before a standardized gluten-free study meal followed approximately 30 minutes later by a standardized 1 gm gluten-containing study meal.
  Interventions: Drug: PvP003 placebo; Drug: PvP003
- Part 4, Cohorts 4A and 4B Healthy Participants (Experimental): Participants will receive multiple dose of PvP003 placebo and 600 mg of PvP003.
  Interventions: Drug: PvP003 placebo; Drug: PvP003
- Part 3, Cohorts 3I and 3J Healthy Participants (Experimental): Participants will receive single dose of PvP003 placebo and 150 mg of PvP003 without pretreatment buffer solution before a standardized 1 gm gluten-containing study meal.
  Interventions: Drug: PvP003 placebo; Drug: PvP003 150 mg

INTERVENTIONS:
Other: PvP001 placebo — placebo
  Arms: Part 1, Cohort 1A-1 to 1D-1 Healthy Participants; Part 1, Cohort 1A-2 - 1D-2 Celiac Disease (CeD); Part 2, Cohort 2A - Cohort 2C Healthy Participants; Part 2, Cohort 2D Healthy Participants; Part 2, Cohort 2F- Cohort 2H Healthy Participants; Part 2, Cohort 2I and Cohort 2J Healthy Participants
Drug: PvP001 100 mg — PvP001 100 mg
  Arms: Part 1, Cohort 1A-1 to 1D-1 Healthy Participants; Part 1, Cohort 1A-2 - 1D-2 Celiac Disease (CeD)
Drug: PvP001 300 mg — PvP001 300 mg
  Arms: Part 1, Cohort 1A-1 to 1D-1 Healthy Participants; Part 1, Cohort 1A-2 - 1D-2 Celiac Disease (CeD); Part 2, Cohort 2F- Cohort 2H Healthy Participants
Drug: PvP001 900 mg — PvP001 900 mg
  Arms: Part 1, Cohort 1A-1 to 1D-1 Healthy Participants; Part 1, Cohort 1A-2 - 1D-2 Celiac Disease (CeD); Part 2, Cohort 2I and Cohort 2J Healthy Participants
Drug: Maximum Feasible Dose (MFD) of PvP002 — MFD of PvP002
  Other Names: MFD of PvP002
  Arms: Part 1, Cohort 1E-1 Healthy Participants; Part 1, Cohort 1E-2 CeD; Part 2, Cohort 2E Healthy Participants
Drug: Maximum Tolerated Dose (MTD) of PvP001 — Maximum Tolerated Dose (MTD) of PvP001
  Arms: Part 2, Cohort 2A - Cohort 2C Healthy Participants; Part 2, Cohort 2D Healthy Participants
Drug: MTD of PvP001 following 7 days of PPI treatment — Maximum Tolerated Dose (MTD) of PvP001 following 7 days of PPI (Proton Pump Inhibitor) treatment
  Arms: Part 2, Cohort 2A - Cohort 2C Healthy Participants
Other: PvP002 placebo — Placebo
  Arms: Part 2, Cohort 2E Healthy Participants
Drug: PvP001 600 mg — PvP001 600 mg
  Arms: Part 2, Cohort 2F- Cohort 2H Healthy Participants
Drug: PvP003 placebo — Placebo tablet orally.
  Arms: Part 3, Cohorts 3A and 3B Healthy Participants; Part 3, Cohorts 3C and 3D Healthy Participants; Part 3, Cohorts 3E and 3F Healthy Participants; Part 3, Cohorts 3G and 3H Healthy Participants; Part 3, Cohorts 3I and 3J Healthy Participants; Part 4, Cohorts 4A and 4B Healthy Participants
Drug: PvP003 — PvP003 tablet orally.
  Arms: Part 3, Cohorts 3A and 3B Healthy Participants; Part 3, Cohorts 3C and 3D Healthy Participants; Part 3, Cohorts 3E and 3F Healthy Participants; Part 3, Cohorts 3G and 3H Healthy Participants; Part 4, Cohorts 4A and 4B Healthy Participants
Drug: PvP003 150 mg — PvP003 150 mg
  Arms: Part 3, Cohorts 3I and 3J Healthy Participants

SUMMARY:
It is hoped that different forms of the same medicine, called PVP001, PVP002, and PVP003, will help people with celiac disease. Both healthy adults and adults with celiac disease will take part in this study.

There are many main aims of the study.

* To check if participants have side effects from different forms of the study medicine. These forms are called PVP001 (liquid in a cup), PVP002 capsule, and PVP003 tablet.
* To check how well PVP003 breaks down gluten.
* To check how much PVP003 participants can take without getting side effects from it.

The study is in 4 parts. At the start of each part of the study, the study doctor will check to determine who can take part at the first study visit. Different groups of participants will be in different parts of the study.

In all parts of the study, some participants will take 1 of the 3 forms of study medicine. Others will take a placebo. In this study, a placebo will look like the form of study medicine but will not have any medicine in it. This means that a placebo can either look like PVP001 liquid in a cup, the PVP002 tablet, or the PVP003 tablet.

In Part 1, different small groups of participants will take lower to higher doses of PVP001 or PVP002 or a placebo. This is to work out the best dose of study medicine to take in other parts of the study. After treatment, participants will regularly visit the clinic to check that they have no problems with their treatment, including any side effects from their treatment.

In Part 2, different small groups will take different doses of PVP001 or PVP002 or a placebo, either with or without a meal that has different amounts of gluten in it. This is to check if PVP001 or PVP002 has broken down gluten in the body. Participants will visit the clinic after treatment to check how much gluten has been broken down in the body.

In Part 3, different small groups will take different doses of PVP003 or a placebo, either with or without a meal that has gluten in it. This is to check if PVP003 has broken down gluten in the body. Participants will visit the clinic after treatment to check if more gluten has broken down in the body.

In Part 4, different small groups will take PVP003 or placebo 3 times a day for 5 days. After treatment, participants will visit the clinic to check that they have no problems with their treatment, including any side effects from their treatment.

DETAILED DESCRIPTION:
This study has four parts. Each part of the study begins with a Screening Period of up to 4 weeks to allow for completion of screening procedures and subject scheduling. Each participant will be screened by means of medical history, medication review, Gastrointestinal Symptoms Questionnaire (GSQ), physical examination, vital signs, weight, height, laboratory tests, and ECG. The GSQ is being used as a separate safety monitoring tool in this study to ensure that all gastrointestinal complaints are reported by the participant.

Following completion of all screening procedures, eligible participants will be enrolled in the study.

Part 1 of the study in healthy participants will be completed prior to enrollment of any subject in Part 2 of the study. A participant enrolled in Part 1 of the study will participate in one of five dose Cohorts. Enrollment of healthy participants and participants with CeD in each of the five dose Cohorts will occur sequentially, but each of these dose Cohorts will be open to enrollment only after demonstration of the safety and tolerability of the same dose level in healthy participants. A healthy participant enrolled in Part 2 of the study will participate in one of three groups; within Groups 1, 2 and 3 enrollment may occur in parallel. A healthy participant enrolled in Part 3 of the study will participate in one of five groups; within Groups 1 to 5 enrollment will occur sequentially. A healthy participant enrolled in Part 4 of the study will participate in two cohorts; enrollment in Part 4 may occur in parallel with enrollment in Part 3. Each participant will be randomized to one of two possible treatment order. Participants who participate in Part 1 or Part 2 of the study, and who are not ADA positive, may participate in Part 3 or Part 4 of the study. No other participants may participate in more than one Part/Group of the study.

ELIGIBILITY:
Inclusion Criteria:

Part 1, Part 2, Part 3 and Part 4

1. Male or female age 18- 64 years, inclusive
2. No relevant gastrointestinal symptoms
3. Able to abstain from alcohol for 72 hours prior to the Screening Visit; for 72 hours prior to and after the Cohort Treatment Day (Part 1, Part 2, and Part 3); for 72 hours prior to the Safety Visit (Part 2 and Part 3); and for 72 hours prior to Day 1 of the first Cohort Treatment Period through the Safety Visit (Part 4).
4. A female participant must have a negative pregnancy test at Screening and on Cohort Treatment Day -1 (Part 1, Part 2, and Part 3) or a negative pregnancy test at Screening and on Day -1 of each Cohort Treatment Period (Part 4), and must agree to continue acceptable birth control measures (example, abstinence, a stable hormonal contraceptive, double-barrier method, or vasectomy in partner) from the Screening Visit through the 28 ± 2 days. Follow Up ADA Blood Sampling Visit
5. A male participant must agree to use acceptable birth control measures (e.g., abstinence, latex condom, or vasectomy), or must have a female partner who will continue birth control measures (e.g., abstinence, a stable hormonal contraceptive, or double-barrier method) from the Screening Visit through the 28 ± 2 days Follow Up Anti-Drug Antibody Blood Sampling Visit
6. Able to read and understand English
7. Able to provide written informed consent

   Additional Inclusion Criteria for Part 1, Part 2, Part 3, and Part 4 Healthy Adult Volunteers
8. No use of over-the-counter or prescription medication, except for birth control medications for the duration of the study
9. No history of gastrointestinal diseases or disorders
10. No history of intolerance, sensitivity, or reactions to gluten or any other food or food ingredient
11. Able to maintain a gluten-free diet for 24 hours prior to the Cohort Treatment Day (Part 1, Part 2, and Part 3), or usually ingests meals three times a day (that is, breakfast, lunch, and dinner) and is able to continue doing so during each Cohort Treatment Period (Part 4)

    Additional Inclusion Criteria for Part 1 Participants with Celiac Disease
12. Documented history of Celiac Disease in medical records
13. Maintaining a gluten-free diet for ≥6 months
14. No use of over-the-counter or prescription medication, except for birth control medications and those allowed by the study doctor, for the duration of the study.
15. No history of gastrointestinal diseases or disorders, other than Celiac Disease
16. No history of intolerance, hypersensitivity, or reaction to any food or food ingredient
17. Able to continue a gluten-free diet for the duration of the study

Exclusion Criteria:

Part 1, Part 2, Part 3, and Part 4

1. Current symptoms or signs of illness
2. Chronic viral infection or immunodeficiency condition
3. Any female who is pregnant, planning to become pregnant during the study, or breast-feeding; any male who is planning to father a child during the study
4. Receipt (or planned receipt) of another investigational medication within 4 weeks prior to the Screening Visit through the duration of the study
5. Alcohol consumption greater than (>) 5 drinks/week, alcohol consumption within 72 hours prior to any study visit (Part 1, Part 2, and Part 3), alcohol consumption within 72 hours prior to Day 1 of the first Cohort Treatment Period through the Safety Visit (Part 4), or a positive alcohol breathalyzer test at any study visit
6. History of illicit or recreational drug use within the three years prior to the Screening Visit, or a positive urine drug screen at any study visit
7. Use of tobacco or nicotine products, including smoking, smokeless tobacco, e-cigarettes, or nicotine replacement products within 12 months prior to the Screening Visit through the duration of the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Pultz IS, Hill M, Vitanza JM, Wolf C, Saaby L, Liu T, Winkle P, Leffler DA. Gluten Degradation, Pharmacokinetics, Safety, and Tolerability of TAK-062, an Engineered Enzyme to Treat Celiac Disease. Gastroenterology. 2021 Jul;161(1):81-93.e3. doi: 10.1053/j.gastro.2021.03.019. Epub 2021 Mar 17. PMID 33741317
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/5fb4db4c17465c002989a1a5

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at 1 investigative site in the United States from 19 June 2018 to 02 July 2021.
Pre-assignment Details: Healthy participants and participants with Celiac Disease (CeD) were enrolled in this 4-part study. In Part 1, healthy participants and participants with CeD were enrolled and in Parts 2, 3 and 4 only healthy participants were enrolled to receive PVP001 (TAK-062 liquid), PVP002 (TAK-062 capsule), and PVP003 (TAK-062 tablet) formulation or matching-placebo.
Groups:
- Part 1, (1A-1): PvP001 Placebo: PvP001 (TAK-062 liquid formulation) placebo-matching liquid, orally, single dose on Cohort Treatment Day in healthy participants.
- Part 1, (1B-1): PvP001 100 mg: PvP001 (TAK-062 liquid formulation) 100 milligram (mg), orally, single dose on Cohort Treatment Day in healthy participants.
- Part 1, (1C-1): PvP001 300 mg: PvP001 (TAK-062 liquid formulation) 300 mg, orally, single dose on Cohort Treatment Day in healthy participants.
- Part 1, (1D-1): PvP001 900 mg: PvP001 (TAK-062 liquid formulation) 900 mg, orally, single dose on Cohort Treatment Day in healthy participants.
- Part 1, (1E-1): PvP002 600 mg: PvP002 (TAK-062 capsule formulation) 600 mg, orally, single dose on Cohort Treatment Day in healthy participants.
- Part 1, (1A-2): PvP001 Placebo: PvP001 (TAK-062 liquid formulation) placebo-matching liquid, orally, single dose on Cohort Treatment Day in CeD participants.
- Part 1, (1B-2): PvP001 100 mg: PvP001 (TAK-062 liquid formulation) 100 mg, orally, single dose on Cohort Treatment Day in CeD participants.
- Part 1, (1C-2): PvP001 300 mg: PvP001 (TAK-062 liquid formulation) 300 mg, orally, single dose on Cohort Treatment Day in CeD participants.
- Part 1, (1D-2): PvP001 900 mg: PvP001 (TAK-062 liquid formulation) 900 mg, orally, single dose on Cohort Treatment Day in CeD participants.
- Part 1, (1E-2): PvP002 600 mg: PvP002 (TAK-062 capsule formulation) 600 mg, orally, single dose on Cohort Treatment Day in CeD participants.
- Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C): PvP001 (TAK-062 liquid formulation) placebo-matching liquid (2A), orally, single dose on Cohort Treatment Day of Cohort 2A, followed by PvP001 900 mg (2B), orally, single dose on Cohort Treatment Day of Cohort 2B, further followed by PvP001 900 mg following 7 days of proton pump inhibitor (PPI) treatment (2C), orally, single dose on Cohort Treatment Day of Cohort 2C in healthy participants. There was a washout period of 7 days between each Cohort Treatment Day.
- Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B): PvP001 (TAK-062 liquid formulation) placebo-matching liquid (2A), orally, single dose on Cohort Treatment Day of Cohort 2A, PvP001 900 mg following 7 days of PPI treatment (2C), orally, single dose on Cohort Treatment Day of Cohort 2C further followed by PvP001 900 mg (2B), orally, single dose on Cohort Treatment Day of Cohort 2B, in healthy participants. There was a washout period of 7 days between each Cohort Treatment Day.
- Part 2, Group 1: PvP001 900 mg (2B) + PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C); Part 2, Group 1: PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A): PvP001 (TAK-062 liquid formulation) 900 mg (2B), orally, single dose on Cohort Treatment Day of Cohort 2B, followed by PvP001 placebo-matching liquid (2A), orally, single dose on Cohort Treatment Day of Cohort 2A, further followed by PvP001 900 mg following 7 days of PPI treatment (2C), orally, single dose on Cohort Treatment Day of Cohort 2C in healthy participants. There was a washout period of 7 days between each Cohort Treatment Day.
- Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) + PvP001 900 mg (2B): PvP001 (TAK-062 liquid formulation) 900 mg following 7 days of PPI treatment (2C), orally, single dose on Cohort Treatment Day of Cohort 2C, followed by PvP001 placebo-matching liquid (2A), orally, single dose on Cohort Treatment Day of Cohort 2A, further followed by PvP001 900 mg (2B), orally, single dose on Cohort Treatment Day of Cohort 2B in healthy participants. There was a washout period of 7 days between each Cohort Treatment Day.
- Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) + PvP001 Placebo (2A): PvP001 (TAK-062 liquid formulation) 900 mg following 7 days of PPI treatment (2C), orally, single dose on Cohort Treatment Day of Cohort 2C, followed by PvP001 900 mg (2B), orally, single dose on Cohort Treatment Day of Cohort 2B, further followed by PvP001 placebo-matching liquid (2A), orally, single dose on Cohort Treatment Day of Cohort 2A in healthy participants. There was a washout period of 7 days between each Cohort Treatment Day.
- Part 2, Group 2: PvP002 Comparator (2D) + PvP002 600 mg (2E): PvP002 capsule comparator (sterile water) (2D), orally, single dose on Cohort Treatment Day of Cohort 2D, followed by PvP002 (TAK-062 capsule formulation) 600 mg (2E), orally, single dose on Cohort Treatment Day of Cohort 2E in healthy participants. There was a washout period of 7 days between each Cohort Treatment Day.
- Part 2, Group 2: PvP002 600 mg (2E) + PvP002 Comparator (2D): PvP002 (TAK-062 capsule formulation) 600 mg (2E), orally, single dose on Cohort Treatment Day of Cohort 2E, followed by PvP002 capsule comparator (sterile water) (2D), orally, single dose on Cohort Treatment Day of Cohort 2D in healthy participants. There was a washout period of 7 days between each Cohort Treatment Day.
- Part 2, Group 3: PvP001 Placebo (2F) + PvP001 300 mg (2G): PvP001 (TAK-062 liquid formulation) placebo-matching liquid (2F), orally, single dose on Cohort Treatment Day of Cohort 2F, followed by PvP001 300 mg (2G), orally, single dose on Cohort Treatment Day of Cohort 2G in healthy participants. There was a washout period of 7 days between each Cohort Treatment Day.
- Part 2, Group 3: PvP001 300 mg (2G) + PvP001 Placebo (2F): PvP001 (TAK-062 liquid formulation) 300 mg (2G), orally, single dose on Cohort Treatment Day of Cohort 2G, followed by PvP001 placebo-matching liquid (2F), orally, single dose on Cohort Treatment Day of Cohort 2F in healthy participants. There was a washout period of 7 days between each Cohort Treatment Day.
- Part 2, Group 3: PvP001 Placebo (2F) + PvP001 600 mg (2H): PvP001 (TAK-062 liquid formulation) placebo-matching liquid (2F), orally, single dose on Cohort Treatment Day of Cohort 2F, followed by PvP001 600 mg (2H), orally, single dose on Cohort Treatment Day of Cohort 2H in healthy participants. There was a washout period of 7 days between each Cohort Treatment Day.
- Part 2, Group 3: PvP001 600 mg (2H) + PvP001 Placebo (2F): PvP001 (TAK-062 liquid formulation) 600 mg (2H), orally, single dose on Cohort Treatment Day of Cohort 2H, followed by PvP001 placebo-matching liquid (2F), orally, single dose on Cohort Treatment Day of Cohort 2F in healthy participants. There was a washout period of 7 days between each Cohort Treatment Day.
- Part 2, Group 3: PvP001 Placebo (2I) + PvP001 900 mg (2J): PvP001 (TAK-062 liquid formulation) placebo-matching liquid (2I), orally, single dose on Cohort Treatment Day of Cohort 2I, followed by PvP001 900 mg (2J), orally, single dose on Cohort Treatment Day of Cohort 2J in healthy participants. There was a washout period of 7 days between each Cohort Treatment Day.
- Part 2, Group 3: PvP001 900 mg (2J) + PvP001 Placebo (2I): PvP001 (TAK-062 liquid formulation) 900 mg (2J), orally, single dose on Cohort Treatment Day of Cohort 2J, followed by PvP001 placebo-matching liquid (2I), orally, single dose on Cohort Treatment Day of Cohort 2I in healthy participants. There was a washout period of 7 days between each Cohort Treatment Day.
- Part 3, Group 1: PvP003 Placebo (3A) + PvP003 600 mg (3B): PvP003 (TAK-062 tablet formulation) placebo-matching tablet (3A) with pretreatment buffer solution administered prior to the PvP003 before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3A, followed by PvP003 600 mg (3B) with pretreatment buffer solution administered prior to the PvP003 before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3B in healthy participants. There was a washout period of 3 days between each Cohort Treatment Day.
- Part 3, Group 1: PvP003 600 mg (3B) + PvP003 Placebo (3A): PvP003 (TAK-062 tablet formulation) 600 mg (3B) with pretreatment buffer solution administered prior to the PvP003 before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3B, followed by PvP003 placebo-matching tablet (3A) with pretreatment buffer solution administered prior to the PvP003 before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3A in healthy participants. There was a washout period of 3 days between each Cohort Treatment Day.
- Part 3, Group 2: PvP003 Placebo (3C) + PvP003 600 mg (3D): PvP003 (TAK-062 tablet formulation) placebo-matching tablet (3C) without pretreatment buffer solution before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3C, followed by PvP003 600 mg (3D) without pretreatment buffer solution before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3D in healthy participants. There was a washout period of 3 days between each Cohort Treatment Day.
- Part 3, Group 2: PvP003 600 mg (3D) + PvP003 Placebo (3C): PvP003 (TAK-062 tablet formulation) 600 mg (3D) without pretreatment buffer solution before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3D, followed by PvP003 placebo-matching tablet (3C) without pretreatment buffer solution before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3C in healthy participants. There was a washout period of 3 days between each Cohort Treatment Day.
- Part 3, Group 3: PvP003 Placebo (3E) + PvP003 600 mg (3F): PvP003 (TAK-062 tablet formulation) placebo-matching tablet (3E) without pretreatment buffer solution administered after an approximately 50 mL portion of standardized 1 gram gluten-containing study meal and then remaining portion of the 1 gram gluten-containing study meal was ingested after administration of PvP0003 orally, single dose on Cohort Treatment Day of Cohort 3E, followed by PvP003 600 mg (3F) without pretreatment buffer solution administered after an approximately 50 mL portion of standardized 1 gram gluten-containing study meal and then remaining portion of the 1 gram gluten-containing study meal was ingested after administration of PvP0003 orally, single dose on Cohort Treatment Day of Cohort 3F in healthy participants. There was a washout period of 3 days between each Cohort Treatment Day.
- Part 3, Group 3: PvP003 600 mg (3F) + PvP003 Placebo (3E): PvP003 (TAK-062 tablet formulation) 600 mg (3F) without pretreatment buffer solution administered after an approximately 50 mL portion of standardized 1 gram gluten-containing study meal and then remaining portion of the 1 gram gluten-containing study meal was ingested after administration of PvP0003 orally, single dose on Cohort Treatment Day of Cohort 3F, followed by PvP003 placebo-matching tablet (3E) without pretreatment buffer solution administered after an approximately 50 mL portion of standardized 1 gram gluten-containing study meal and then remaining portion of the 1 gram gluten-containing study meal was ingested after administration of PvP0003, orally, single dose on Cohort Treatment Day of Cohort 3E, in healthy participants. There was a washout period of 3 days between each Cohort Treatment Day.
- Part 3, Group 4: PvP003 Placebo (3G) + PvP003 600 mg (3H): PvP003 (TAK-062 tablet formulation) placebo-matching tablet (3G) without pretreatment buffer solution before standardized gluten-free study meal followed by a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3G, followed by PvP003 600 mg (3H) without pretreatment buffer solution before standardized gluten-free study meal followed by a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3H in healthy participants. There was a washout period of 3 days between each Cohort Treatment Day.
- Part 3, Group 4: PvP003 600 mg (3H) + PvP003 Placebo (3G): PvP003 (TAK-062 tablet formulation) 600 mg (3H) without pretreatment buffer solution before standardized gluten-free study meal followed by a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3H, followed by PvP003 placebo-matching tablet (3G) without pretreatment buffer solution before standardized gluten-free study meal followed by a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3G, in healthy participants. There was a washout period of 3 days between each Cohort Treatment Day.
- Part 3, Group 5: PvP003 Placebo (3I) + PvP003 150 mg (3J): PvP003 (TAK-062 tablet formulation) placebo-matching tablet (3I) without pretreatment buffer solution before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3I, followed by PvP003 150 mg (3J) without pretreatment buffer solution before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3J in healthy participants. There was a washout period of 3 days between each Cohort Treatment Day.
- Part 3, Group 5: PvP003 150 mg (3J) + PvP003 Placebo (3I): PvP003 (TAK-062 tablet formulation) 150 mg (3J) without pretreatment buffer solution before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3J, followed by PvP003 placebo-matching tablet (3I) without pretreatment buffer solution before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3I in healthy participants. There was a washout period of 3 days between each Cohort Treatment Day.
- Part 4: PvP003 Placebo, TID (4A) + PvP003 600 mg, TID (4B): PvP003 (TAK-062 tablet formulation) placebo-matching tablet, administered as two tablets of PvP003 placebo, orally, thrice a day (TID) on Treatment Days 1 to 5 (4A) of Cohort Treatment Period 1, followed by PvP003 600 mg administered as two tablets of PvP003 300 mg, orally, TID on Treatment Days 1 to 5 (4B) of Cohort Treatment Period 2 in healthy participants. There was a washout period of 3 days between the two Cohort Treatment Periods.
- Part 4: PvP003 600 mg, TID (4B) + PvP003 Placebo, TID (4A): PvP003 (TAK-062 tablet formulation) 600 mg, administered as two tablets of PvP003 300 mg, orally, TID on Treatment Days 1 to 5 (4B) of Cohort Treatment Period 1, followed by PvP003 placebo-matching tablet, administered as two tablets of PvP003 placebo, orally, TID on Treatment Days 1 to 5 (4A) of Cohort Treatment Period 2 in healthy participants. There was a washout period of 3 days between the two Cohort Treatment Periods.
Period: Part 1 (Day 1)
Arm/Group | Part 1, (1A-1): PvP001 Placebo | Part 1, (1B-1): PvP001 100 mg | Part 1, (1C-1): PvP001 300 mg | Part 1, (1D-1): PvP001 900 mg | Part 1, (1E-1): PvP002 600 mg | Part 1, (1A-2): PvP001 Placebo | Part 1, (1B-2): PvP001 100 mg | Part 1, (1C-2): PvP001 300 mg | Part 1, (1D-2): PvP001 900 mg | Part 1, (1E-2): PvP002 600 mg | Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) | Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg (2B) + PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) | Part 2, Group 1: PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) | Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) + PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) + PvP001 Placebo (2A) | Part 2, Group 2: PvP002 Comparator (2D) + PvP002 600 mg (2E) | Part 2, Group 2: PvP002 600 mg (2E) + PvP002 Comparator (2D) | Part 2, Group 3: PvP001 Placebo (2F) + PvP001 300 mg (2G) | Part 2, Group 3: PvP001 300 mg (2G) + PvP001 Placebo (2F) | Part 2, Group 3: PvP001 Placebo (2F) + PvP001 600 mg (2H) | Part 2, Group 3: PvP001 600 mg (2H) + PvP001 Placebo (2F) | Part 2, Group 3: PvP001 Placebo (2I) + PvP001 900 mg (2J) | Part 2, Group 3: PvP001 900 mg (2J) + PvP001 Placebo (2I) | Part 3, Group 1: PvP003 Placebo (3A) + PvP003 600 mg (3B) | Part 3, Group 1: PvP003 600 mg (3B) + PvP003 Placebo (3A) | Part 3, Group 2: PvP003 Placebo (3C) + PvP003 600 mg (3D) | Part 3, Group 2: PvP003 600 mg (3D) + PvP003 Placebo (3C) | Part 3, Group 3: PvP003 Placebo (3E) + PvP003 600 mg (3F) | Part 3, Group 3: PvP003 600 mg (3F) + PvP003 Placebo (3E) | Part 3, Group 4: PvP003 Placebo (3G) + PvP003 600 mg (3H) | Part 3, Group 4: PvP003 600 mg (3H) + PvP003 Placebo (3G) | Part 3, Group 5: PvP003 Placebo (3I) + PvP003 150 mg (3J) | Part 3, Group 5: PvP003 150 mg (3J) + PvP003 Placebo (3I) | Part 4: PvP003 Placebo, TID (4A) + PvP003 600 mg, TID (4B) | Part 4: PvP003 600 mg, TID (4B) + PvP003 Placebo, TID (4A)
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Day 1)
Arm/Group | Part 1, (1A-1): PvP001 Placebo | Part 1, (1B-1): PvP001 100 mg | Part 1, (1C-1): PvP001 300 mg | Part 1, (1D-1): PvP001 900 mg | Part 1, (1E-1): PvP002 600 mg | Part 1, (1A-2): PvP001 Placebo | Part 1, (1B-2): PvP001 100 mg | Part 1, (1C-2): PvP001 300 mg | Part 1, (1D-2): PvP001 900 mg | Part 1, (1E-2): PvP002 600 mg | Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) | Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg (2B) + PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) | Part 2, Group 1: PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) | Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) + PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) + PvP001 Placebo (2A) | Part 2, Group 2: PvP002 Comparator (2D) + PvP002 600 mg (2E) | Part 2, Group 2: PvP002 600 mg (2E) + PvP002 Comparator (2D) | Part 2, Group 3: PvP001 Placebo (2F) + PvP001 300 mg (2G) | Part 2, Group 3: PvP001 300 mg (2G) + PvP001 Placebo (2F) | Part 2, Group 3: PvP001 Placebo (2F) + PvP001 600 mg (2H) | Part 2, Group 3: PvP001 600 mg (2H) + PvP001 Placebo (2F) | Part 2, Group 3: PvP001 Placebo (2I) + PvP001 900 mg (2J) | Part 2, Group 3: PvP001 900 mg (2J) + PvP001 Placebo (2I) | Part 3, Group 1: PvP003 Placebo (3A) + PvP003 600 mg (3B) | Part 3, Group 1: PvP003 600 mg (3B) + PvP003 Placebo (3A) | Part 3, Group 2: PvP003 Placebo (3C) + PvP003 600 mg (3D) | Part 3, Group 2: PvP003 600 mg (3D) + PvP003 Placebo (3C) | Part 3, Group 3: PvP003 Placebo (3E) + PvP003 600 mg (3F) | Part 3, Group 3: PvP003 600 mg (3F) + PvP003 Placebo (3E) | Part 3, Group 4: PvP003 Placebo (3G) + PvP003 600 mg (3H) | Part 3, Group 4: PvP003 600 mg (3H) + PvP003 Placebo (3G) | Part 3, Group 5: PvP003 Placebo (3I) + PvP003 150 mg (3J) | Part 3, Group 5: PvP003 150 mg (3J) + PvP003 Placebo (3I) | Part 4: PvP003 Placebo, TID (4A) + PvP003 600 mg, TID (4B) | Part 4: PvP003 600 mg, TID (4B) + PvP003 Placebo, TID (4A)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3 | 2 | 3 | 2 | 4 | 7 | 7 | 4 | 4 | 4 | 4 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1 | 2 | 2 | 4 | 5 | 4 | 4 | 4 | 3 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 0 | 2 | 3 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject Non-compliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3 (Day 1)
Arm/Group | Part 1, (1A-1): PvP001 Placebo | Part 1, (1B-1): PvP001 100 mg | Part 1, (1C-1): PvP001 300 mg | Part 1, (1D-1): PvP001 900 mg | Part 1, (1E-1): PvP002 600 mg | Part 1, (1A-2): PvP001 Placebo | Part 1, (1B-2): PvP001 100 mg | Part 1, (1C-2): PvP001 300 mg | Part 1, (1D-2): PvP001 900 mg | Part 1, (1E-2): PvP002 600 mg | Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) | Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg (2B) + PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) | Part 2, Group 1: PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) | Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) + PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) + PvP001 Placebo (2A) | Part 2, Group 2: PvP002 Comparator (2D) + PvP002 600 mg (2E) | Part 2, Group 2: PvP002 600 mg (2E) + PvP002 Comparator (2D) | Part 2, Group 3: PvP001 Placebo (2F) + PvP001 300 mg (2G) | Part 2, Group 3: PvP001 300 mg (2G) + PvP001 Placebo (2F) | Part 2, Group 3: PvP001 Placebo (2F) + PvP001 600 mg (2H) | Part 2, Group 3: PvP001 600 mg (2H) + PvP001 Placebo (2F) | Part 2, Group 3: PvP001 Placebo (2I) + PvP001 900 mg (2J) | Part 2, Group 3: PvP001 900 mg (2J) + PvP001 Placebo (2I) | Part 3, Group 1: PvP003 Placebo (3A) + PvP003 600 mg (3B) | Part 3, Group 1: PvP003 600 mg (3B) + PvP003 Placebo (3A) | Part 3, Group 2: PvP003 Placebo (3C) + PvP003 600 mg (3D) | Part 3, Group 2: PvP003 600 mg (3D) + PvP003 Placebo (3C) | Part 3, Group 3: PvP003 Placebo (3E) + PvP003 600 mg (3F) | Part 3, Group 3: PvP003 600 mg (3F) + PvP003 Placebo (3E) | Part 3, Group 4: PvP003 Placebo (3G) + PvP003 600 mg (3H) | Part 3, Group 4: PvP003 600 mg (3H) + PvP003 Placebo (3G) | Part 3, Group 5: PvP003 Placebo (3I) + PvP003 150 mg (3J) | Part 3, Group 5: PvP003 150 mg (3J) + PvP003 Placebo (3I) | Part 4: PvP003 Placebo, TID (4A) + PvP003 600 mg, TID (4B) | Part 4: PvP003 600 mg, TID (4B) + PvP003 Placebo, TID (4A)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 2 | 5 | 3 | 4 | 4 | 6 | 7 | 9 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 1 | 5 | 3 | 2 | 3 | 3 | 5 | 7 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 3 | 2 | 2 | 0 | 0
Not completed — Subject Non-compliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Subject Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Period: Part 4, Period 1 (Days 1 to 5)
Arm/Group | Part 1, (1A-1): PvP001 Placebo | Part 1, (1B-1): PvP001 100 mg | Part 1, (1C-1): PvP001 300 mg | Part 1, (1D-1): PvP001 900 mg | Part 1, (1E-1): PvP002 600 mg | Part 1, (1A-2): PvP001 Placebo | Part 1, (1B-2): PvP001 100 mg | Part 1, (1C-2): PvP001 300 mg | Part 1, (1D-2): PvP001 900 mg | Part 1, (1E-2): PvP002 600 mg | Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) | Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg (2B) + PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) | Part 2, Group 1: PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) | Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) + PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) + PvP001 Placebo (2A) | Part 2, Group 2: PvP002 Comparator (2D) + PvP002 600 mg (2E) | Part 2, Group 2: PvP002 600 mg (2E) + PvP002 Comparator (2D) | Part 2, Group 3: PvP001 Placebo (2F) + PvP001 300 mg (2G) | Part 2, Group 3: PvP001 300 mg (2G) + PvP001 Placebo (2F) | Part 2, Group 3: PvP001 Placebo (2F) + PvP001 600 mg (2H) | Part 2, Group 3: PvP001 600 mg (2H) + PvP001 Placebo (2F) | Part 2, Group 3: PvP001 Placebo (2I) + PvP001 900 mg (2J) | Part 2, Group 3: PvP001 900 mg (2J) + PvP001 Placebo (2I) | Part 3, Group 1: PvP003 Placebo (3A) + PvP003 600 mg (3B) | Part 3, Group 1: PvP003 600 mg (3B) + PvP003 Placebo (3A) | Part 3, Group 2: PvP003 Placebo (3C) + PvP003 600 mg (3D) | Part 3, Group 2: PvP003 600 mg (3D) + PvP003 Placebo (3C) | Part 3, Group 3: PvP003 Placebo (3E) + PvP003 600 mg (3F) | Part 3, Group 3: PvP003 600 mg (3F) + PvP003 Placebo (3E) | Part 3, Group 4: PvP003 Placebo (3G) + PvP003 600 mg (3H) | Part 3, Group 4: PvP003 600 mg (3H) + PvP003 Placebo (3G) | Part 3, Group 5: PvP003 Placebo (3I) + PvP003 150 mg (3J) | Part 3, Group 5: PvP003 150 mg (3J) + PvP003 Placebo (3I) | Part 4: PvP003 Placebo, TID (4A) + PvP003 600 mg, TID (4B) | Part 4: PvP003 600 mg, TID (4B) + PvP003 Placebo, TID (4A)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 (Part 4 had crossover-design where participants were enrolled in Cohort Treatment Period 1, and entered the Cohort Treatment Period 2 after 3 days of washout period.) | 3 (Part 4 had crossover-design where participants were enrolled in Cohort Treatment Period 1, and entered the Cohort Treatment Period 2 after 3 days of washout period.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 4, Washout Period (3 Days)
Arm/Group | Part 1, (1A-1): PvP001 Placebo | Part 1, (1B-1): PvP001 100 mg | Part 1, (1C-1): PvP001 300 mg | Part 1, (1D-1): PvP001 900 mg | Part 1, (1E-1): PvP002 600 mg | Part 1, (1A-2): PvP001 Placebo | Part 1, (1B-2): PvP001 100 mg | Part 1, (1C-2): PvP001 300 mg | Part 1, (1D-2): PvP001 900 mg | Part 1, (1E-2): PvP002 600 mg | Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) | Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg (2B) + PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) | Part 2, Group 1: PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) | Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) + PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) + PvP001 Placebo (2A) | Part 2, Group 2: PvP002 Comparator (2D) + PvP002 600 mg (2E) | Part 2, Group 2: PvP002 600 mg (2E) + PvP002 Comparator (2D) | Part 2, Group 3: PvP001 Placebo (2F) + PvP001 300 mg (2G) | Part 2, Group 3: PvP001 300 mg (2G) + PvP001 Placebo (2F) | Part 2, Group 3: PvP001 Placebo (2F) + PvP001 600 mg (2H) | Part 2, Group 3: PvP001 600 mg (2H) + PvP001 Placebo (2F) | Part 2, Group 3: PvP001 Placebo (2I) + PvP001 900 mg (2J) | Part 2, Group 3: PvP001 900 mg (2J) + PvP001 Placebo (2I) | Part 3, Group 1: PvP003 Placebo (3A) + PvP003 600 mg (3B) | Part 3, Group 1: PvP003 600 mg (3B) + PvP003 Placebo (3A) | Part 3, Group 2: PvP003 Placebo (3C) + PvP003 600 mg (3D) | Part 3, Group 2: PvP003 600 mg (3D) + PvP003 Placebo (3C) | Part 3, Group 3: PvP003 Placebo (3E) + PvP003 600 mg (3F) | Part 3, Group 3: PvP003 600 mg (3F) + PvP003 Placebo (3E) | Part 3, Group 4: PvP003 Placebo (3G) + PvP003 600 mg (3H) | Part 3, Group 4: PvP003 600 mg (3H) + PvP003 Placebo (3G) | Part 3, Group 5: PvP003 Placebo (3I) + PvP003 150 mg (3J) | Part 3, Group 5: PvP003 150 mg (3J) + PvP003 Placebo (3I) | Part 4: PvP003 Placebo, TID (4A) + PvP003 600 mg, TID (4B) | Part 4: PvP003 600 mg, TID (4B) + PvP003 Placebo, TID (4A)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 4, Period 2 (Days 1 to 5)
Arm/Group | Part 1, (1A-1): PvP001 Placebo | Part 1, (1B-1): PvP001 100 mg | Part 1, (1C-1): PvP001 300 mg | Part 1, (1D-1): PvP001 900 mg | Part 1, (1E-1): PvP002 600 mg | Part 1, (1A-2): PvP001 Placebo | Part 1, (1B-2): PvP001 100 mg | Part 1, (1C-2): PvP001 300 mg | Part 1, (1D-2): PvP001 900 mg | Part 1, (1E-2): PvP002 600 mg | Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) | Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg (2B) + PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) | Part 2, Group 1: PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) | Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) + PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) + PvP001 Placebo (2A) | Part 2, Group 2: PvP002 Comparator (2D) + PvP002 600 mg (2E) | Part 2, Group 2: PvP002 600 mg (2E) + PvP002 Comparator (2D) | Part 2, Group 3: PvP001 Placebo (2F) + PvP001 300 mg (2G) | Part 2, Group 3: PvP001 300 mg (2G) + PvP001 Placebo (2F) | Part 2, Group 3: PvP001 Placebo (2F) + PvP001 600 mg (2H) | Part 2, Group 3: PvP001 600 mg (2H) + PvP001 Placebo (2F) | Part 2, Group 3: PvP001 Placebo (2I) + PvP001 900 mg (2J) | Part 2, Group 3: PvP001 900 mg (2J) + PvP001 Placebo (2I) | Part 3, Group 1: PvP003 Placebo (3A) + PvP003 600 mg (3B) | Part 3, Group 1: PvP003 600 mg (3B) + PvP003 Placebo (3A) | Part 3, Group 2: PvP003 Placebo (3C) + PvP003 600 mg (3D) | Part 3, Group 2: PvP003 600 mg (3D) + PvP003 Placebo (3C) | Part 3, Group 3: PvP003 Placebo (3E) + PvP003 600 mg (3F) | Part 3, Group 3: PvP003 600 mg (3F) + PvP003 Placebo (3E) | Part 3, Group 4: PvP003 Placebo (3G) + PvP003 600 mg (3H) | Part 3, Group 4: PvP003 600 mg (3H) + PvP003 Placebo (3G) | Part 3, Group 5: PvP003 Placebo (3I) + PvP003 150 mg (3J) | Part 3, Group 5: PvP003 150 mg (3J) + PvP003 Placebo (3I) | Part 4: PvP003 Placebo, TID (4A) + PvP003 600 mg, TID (4B) | Part 4: PvP003 600 mg, TID (4B) + PvP003 Placebo, TID (4A)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of study drug.
Groups:
- Part 1, (1B-1): PvP001 100 mg: PvP001 (TAK-062 liquid formulation) 100 mg, orally, single dose on Cohort Treatment Day in healthy participants.
- Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C): PvP001 (TAK-062 liquid formulation) placebo-matching liquid (2A), orally, single dose on Cohort Treatment Day of Cohort 2A, followed by PvP001 900 mg (2B), orally, single dose on Cohort Treatment Day of Cohort 2B, further followed by PvP001 900 mg following 7 days of PPI treatment (2C), orally, single dose on Cohort Treatment Day of Cohort 2C in healthy participants. There was a washout period of 7 days between each Cohort Treatment Day.
- Part 4: PvP003 Placebo, TID (4A) + PvP003 600 mg, TID (4B): PvP003 (TAK-062 tablet formulation) placebo-matching tablet, administered as two tablets of PvP003 placebo, orally, TID on Treatment Days 1 to 5 (4A) of Cohort Treatment Period 1, followed by PvP003 600 mg administered as two tablets of PvP003 300 mg, orally, TID on Treatment Days 1 to 5 (4B) of Cohort Treatment Period 2 in healthy participants. There was a washout period of 3 days between the two Cohort Treatment Periods.
- Total: Total of all reporting groups
Arm/Group | Part 1, (1A-1): PvP001 Placebo | Part 1, (1B-1): PvP001 100 mg | Part 1, (1C-1): PvP001 300 mg | Part 1, (1D-1): PvP001 900 mg | Part 1, (1E-1): PvP002 600 mg | Part 1, (1A-2): PvP001 Placebo | Part 1, (1B-2): PvP001 100 mg | Part 1, (1C-2): PvP001 300 mg | Part 1, (1D-2): PvP001 900 mg | Part 1, (1E-2): PvP002 600 mg | Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) | Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg (2B) + PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) | Part 2, Group 1: PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) | Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) + PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) + PvP001 Placebo (2A) | Part 2, Group 2: PvP002 Comparator (2D) + PvP002 600 mg (2E) | Part 2, Group 2: PvP002 600 mg (2E) + PvP002 Comparator (2D) | Part 2, Group 3: PvP001 Placebo (2F) + PvP001 300 mg (2G) | Part 2, Group 3: PvP001 300 mg (2G) + PvP001 Placebo (2F) | Part 2, Group 3: PvP001 Placebo (2F) + PvP001 600 mg (2H) | Part 2, Group 3: PvP001 600 mg (2H) + PvP001 Placebo (2F) | Part 2, Group 3: PvP001 Placebo (2I) + PvP001 900 mg (2J) | Part 2, Group 3: PvP001 900 mg (2J) + PvP001 Placebo (2I) | Part 3, Group 1: PvP003 Placebo (3A) + PvP003 600 mg (3B) | Part 3, Group 1: PvP003 600 mg (3B) + PvP003 Placebo (3A) | Part 3, Group 2: PvP003 Placebo (3C) + PvP003 600 mg (3D) | Part 3, Group 2: PvP003 600 mg (3D) + PvP003 Placebo (3C) | Part 3, Group 3: PvP003 Placebo (3E) + PvP003 600 mg (3F) | Part 3, Group 3: PvP003 600 mg (3F) + PvP003 Placebo (3E) | Part 3, Group 4: PvP003 Placebo (3G) + PvP003 600 mg (3H) | Part 3, Group 4: PvP003 600 mg (3H) + PvP003 Placebo (3G) | Part 3, Group 5: PvP003 Placebo (3I) + PvP003 150 mg (3J) | Part 3, Group 5: PvP003 150 mg (3J) + PvP003 Placebo (3I) | Part 4: PvP003 Placebo, TID (4A) + PvP003 600 mg, TID (4B) | Part 4: PvP003 600 mg, TID (4B) + PvP003 Placebo, TID (4A) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 1 | 3 | 3 | 2 | 2 | 2 | 2 | 4 | 5 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 4 | 1 | 5 | 3 | 3 | 3 | 3 | 5 | 8 | 3 | 3 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 1 | 3 | 3 | 2 | 2 | 2 | 2 | 4 | 5 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 4 | 1 | 5 | 3 | 3 | 3 | 3 | 5 | 8 | 3 | 3 | 119
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 0 | 2 | 1 | 2 | 1 | 3 | 1 | 1 | 3 | 2 | 0 | 1 | 1 | 2 | 2 | 0 | 1 | 44
  Male | 3 | 3 | 2 | 3 | 3 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 2 | 2 | 2 | 2 | 3 | 2 | 1 | 4 | 2 | 3 | 2 | 3 | 0 | 3 | 0 | 2 | 1 | 3 | 2 | 2 | 3 | 6 | 3 | 2 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 0 | 3 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 3 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 2 | 2 | 2 | 0 | 33
  Not Hispanic or Latino | 3 | 2 | 3 | 2 | 3 | 0 | 1 | 2 | 3 | 1 | 2 | 3 | 1 | 1 | 1 | 2 | 4 | 3 | 1 | 4 | 3 | 4 | 2 | 3 | 3 | 3 | 1 | 3 | 2 | 3 | 2 | 2 | 3 | 6 | 1 | 3 | 86
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 2 | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 2 | 4 | 1 | 0 | 32
  White | 0 | 2 | 0 | 1 | 3 | 3 | 3 | 3 | 3 | 1 | 2 | 1 | 0 | 2 | 2 | 1 | 2 | 3 | 4 | 3 | 2 | 3 | 3 | 2 | 1 | 3 | 0 | 5 | 2 | 2 | 1 | 2 | 3 | 3 | 2 | 2 | 75
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 1 | 3 | 3 | 2 | 2 | 2 | 2 | 4 | 5 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 4 | 1 | 5 | 3 | 3 | 3 | 3 | 5 | 8 | 3 | 3 | 119

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants Reporting One or More Treatment Emergent Adverse Events (TEAEs) for PvP001 and PvP002
Time Frame: Cohort Treatment Day up to 5 days after 24-hour safety assessment on Day 2 (up to Day 7)
Population: Safety population included all participants who received at least one dose of study drug. As planned, this outcome measure was assessed only for Part 1 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, (1A-1): PvP001 Placebo | Part 1, (1B-1): PvP001 100 mg | Part 1, (1C-1): PvP001 300 mg | Part 1, (1D-1): PvP001 900 mg | Part 1, (1E-1): PvP002 600 mg | Part 1, (1A-2): PvP001 Placebo | Part 1, (1B-2): PvP001 100 mg | Part 1, (1C-2): PvP001 300 mg | Part 1, (1D-2): PvP001 900 mg | Part 1, (1E-2): PvP002 600 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 1

2. Primary Outcome: Part 4: Number of Participants Reporting One or More TEAEs for PvP003 After Multiple Doses
Time Frame: Day 1 of Cohort Treatment Period 1 up to 5 days after the Day 5 of Cohort Treatment Period 2 (up to Day 28)
Population: Safety population included all participants who received at least one dose of study drug. As planned, this outcome measure was assessed only for Part 4 of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Part 4: PvP003 Placebo, TID (4A): PvP003 (TAK-062 tablet formulation) placebo-matching tablet, administered as two tablets of PvP003 placebo, orally, TID on Treatment Days 1 to 5 (4A) of Cohort Treatment Period 1 or 2 in healthy participants.
- Part 4: PvP003 600 mg, TID (4B): PvP003 (TAK-062 tablet formulation) 600 mg, administered as two tablets of PvP003 300 mg, orally, TID on Treatment Days 1 to 5 (4B) of Cohort Treatment Period 1 or 2 in healthy participants.
Arm/Group | Part 4: PvP003 Placebo, TID (4A) | Part 4: PvP003 600 mg, TID (4B)
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

3. Primary Outcome: Part 1: Number of Participants Reporting One or More Treatment Emergent Serious Adverse Events (TESAEs) for PvP001 and PvP002
Time Frame: Cohort Treatment Day up to 5 days after 24-hour safety assessment on Day 2 (up to Day 7)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, (1A-1): PvP001 Placebo | Part 1, (1B-1): PvP001 100 mg | Part 1, (1C-1): PvP001 300 mg | Part 1, (1D-1): PvP001 900 mg | Part 1, (1E-1): PvP002 600 mg | Part 1, (1A-2): PvP001 Placebo | Part 1, (1B-2): PvP001 100 mg | Part 1, (1C-2): PvP001 300 mg | Part 1, (1D-2): PvP001 900 mg | Part 1, (1E-2): PvP002 600 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part 4: Number of Participants Reporting One or More TESAEs for PvP003 600 mg After Multiple Doses
Time Frame: Day 1 of Cohort Treatment Period 1 up to 5 days after the Day 5 of Cohort Treatment Period 2 (up to Day 28)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 4: PvP003 Placebo, TID (4A) | Part 4: PvP003 600 mg, TID (4B)
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

5. Primary Outcome: Part 2, Group 1, Cohort 2B: Median Percentage of Gluten Degradation by PvP001 in a Standardized 3 Gram (gm) Gluten-containing Study Meal After Administration of PvP001
Description: Median percentage degraded relative to placebo was derived using the formula: (1 - [active/placebo])*100. Gluten degradation was assessed using Enzyme-Linked Immunosorbent Assay (ELISA) based on the monoclonal R5 and G12 antibodies.
Time Frame: Cohort Treatment Day
Population: Intent-to-Treat (ITT) population in Part 2 of the study, included all participants who received at least one dose of study drug. As planned, this outcome measure was assessed in Group 1, Cohort 2B (PvP001 900 mg) of Part 2 only. Here 'N' (overall number of participants analyzed) included all participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: percentage of gluten degradation
Groups:
- Part 2, Group 1: PvP001 900 mg (2B): PvP001 (TAK-062 liquid formulation) 900 mg (2B), orally, single dose on Cohort Treatment Day of Cohort 2B in healthy participants.
Arm/Group | Part 2, Group 1: PvP001 900 mg (2B)
Number analyzed (Participants) | 11
percentage of gluten degradation
  R5 | 94.41 [79.7 to 99.9]
  G12 | 97.89 [79.6 to 99.9]

6. Primary Outcome: Part 2, Group 2, Cohort 2E: Median Percentage of Gluten Degradation by PvP002 in a Standardized 3 gm Gluten-containing Study Meal After Administration of PvP002
Description: Median percentage degraded relative to placebo was derived using the formula: (1 - [active/placebo])*100. Gluten degradation was assessed using ELISA based on the monoclonal R5 and G12 antibodies.
Time Frame: Cohort Treatment Day
Population: ITT population in Part 2 of the study, included all participants who received at least one dose of study drug. As planned, this outcome measure was assessed in Group 2, Cohort 2E (PvP002 600 mg) of Part 2 only. Here 'N' (overall number of participants analyzed) included all participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: percentage of gluten degradation
Groups:
- Part 2, Group 2: PvP002 600 mg (2E): PvP002 (TAK-062 capsule formulation) 600 mg (2E), orally, single dose on Cohort Treatment Day of Cohort 2E in healthy participants.
Arm/Group | Part 2, Group 2: PvP002 600 mg (2E)
Number analyzed (Participants) | 9
percentage of gluten degradation
  R5 | 99.67 [0.0 to 99.8]
  G12 | 99.70 [0.0 to 99.9]

7. Primary Outcome: Part 2, Group 1, Cohort 2C: Median Percentage of Gluten Degradation by PvP001 in a Standardized 3 gm Gluten-containing Study Meal Following 7 Days of Standard Dose PPI Treatment
Description: as for outcome 6
Time Frame: Cohort Treatment Day
Population: ITT population in Part 2 of the study, included all participants who received at least one dose of study drug. As planned, this outcome measure was assessed in Group 1, Cohort 2C (PvP001 900 mg) of Part 2 only. Here 'N' (overall number of participants analyzed) included all participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: percentage of gluten degradation
Groups:
- Part 2, Group 1: PvP001 900 mg With PPI (2C): PvP001 (TAK-062 liquid formulation) 900 mg following 7 days of PPI treatment (2C), orally, single dose on Cohort Treatment Day of Cohort 2C in healthy participants.
Arm/Group | Part 2, Group 1: PvP001 900 mg With PPI (2C)
Number analyzed (Participants) | 12
percentage of gluten degradation
  R5 | 99.44 [92.3 to 99.9]
  G12 | 99.62 [97.6 to 99.8]

8. Primary Outcome: Part 2, Group 3, Cohort 2G and 2H: Median Percentage of Gluten Degradation by PvP001 300 mg and 600 mg in a Standardized 1 gm Gluten-containing Study Meal at 20 Minutes After Administration of PvP001
Description: as for outcome 6
Time Frame: Cohort Treatment Day: at 20 minutes post-dose
Population: ITT population in Part 2 of the study, included all participants who received at least one dose of study drug. As planned, this outcome measure was assessed in Group 3, Cohort 2G (PvP001 300 mg) and Cohort 2H (PvP001 600 mg) of Part 2 only.
Measure: Median (Full Range); unit: percentage of gluten degradation
Groups:
- Part 2, Group 3: PvP001 300 mg (2G): PvP001 (TAK-062 liquid formulation) 300 mg (2G), orally, single dose on Cohort Treatment Day of Cohort 2G in healthy participants.
- Part 2, Group 3: PvP001 600 mg (2H): PvP001 (TAK-062 liquid formulation) 600 mg (2H), orally, single dose on Cohort Treatment Day of Cohort 2H in healthy participants.
Arm/Group | Part 2, Group 3: PvP001 300 mg (2G) | Part 2, Group 3: PvP001 600 mg (2H)
Number analyzed (Participants) | 8 | 8
percentage of gluten degradation
  R5: 20 minutes | 95.89 [55.6 to 99.2] | 98.13 [95.0 to 99.9]
  G12: 20 minutes | 97.63 [85.3 to 99.3] | 97.98 [89.2 to 99.9]

9. Primary Outcome: Part 2, Group 3, Cohort 2G and 2H: Median Percentage of Gluten Degradation by PvP001 300 mg and 600 mg in a Standardized 1 gm Gluten-containing Study Meal at 35 Minutes After Administration of PvP001
Description: as for outcome 6
Time Frame: Cohort Treatment Day: at 35 minutes post-dose
Population: as for outcome 8
Measure: Median (Full Range); unit: percentage of gluten degradation
Arm/Group | Part 2, Group 3: PvP001 300 mg (2G) | Part 2, Group 3: PvP001 600 mg (2H)
Number analyzed (Participants) | 8 | 8
percentage of gluten degradation
  R5: 35 minutes | 98.19 [87.9 to 99.6] | 98.95 [84.1 to 99.9]
  G12: 35 minutes | 97.92 [93.9 to 99.6] | 98.43 [60.3 to 99.9]

10. Primary Outcome: Part 2, Group 3, Cohort 2G and 2H: Median Percentage of Gluten Degradation by PvP001 300 mg and 600 mg in a Standardized 1 gm Gluten-containing Study Meal at 65 Minutes After Administration of PvP001
Description: as for outcome 6
Time Frame: Cohort Treatment Day: at 65 minutes post-dose
Population: as for outcome 8
Measure: Median (Full Range); unit: percentage of gluten degradation
Arm/Group | Part 2, Group 3: PvP001 300 mg (2G) | Part 2, Group 3: PvP001 600 mg (2H)
Number analyzed (Participants) | 8 | 8
percentage of gluten degradation
  R5: 65 minutes | 95.21 [83.8 to 98.4] | 98.15 [85.6 to 99.9]
  G12: 65 minutes | 96.30 [86.8 to 99.5] | 98.87 [82.1 to 99.9]

11. Primary Outcome: Part 2, Group 3, Cohort 2J: Median Percentage of Gluten Degradation by PvP001 900 mg in a Standardized 6 gm Gluten-containing Study Meal at 20 Minutes After Administration of PvP001
Description: as for outcome 6
Time Frame: Cohort Treatment Day: at 20 minutes post-dose
Population: ITT population in Part 2 of the study, included all participants who received at least one dose of study drug. As planned, this outcome measure was assessed in Group 3, Cohort 2J (PvP001 900 mg) of Part 2 only.
Measure: Median (Full Range); unit: percentage of gluten degradation
Groups:
- Part 2, Group 3: PvP001 900 mg (2J): PvP001 (TAK-062 liquid formulation) 900 mg (2J), orally, single dose on Cohort Treatment Day of Cohort 2J in healthy participants.
Arm/Group | Part 2, Group 3: PvP001 900 mg (2J)
Number analyzed (Participants) | 8
percentage of gluten degradation
  R5: 20 minutes | 99.82 [62.2 to 100.0]
  G12: 20 minutes | 99.77 [85.2 to 99.9]

12. Primary Outcome: Part 2, Group 3, Cohort 2J: Median Percentage of Gluten Degradation by PvP001 900 mg in a Standardized 6 gm Gluten-containing Study Meal at 35 Minutes After Administration of PvP001
Description: as for outcome 6
Time Frame: Cohort Treatment Day: at 35 minutes post-dose
Population: as for outcome 11
Measure: Median (Full Range); unit: percentage of gluten degradation
Arm/Group | Part 2, Group 3: PvP001 900 mg (2J)
Number analyzed (Participants) | 8
percentage of gluten degradation
  R5: 35 minutes | 99.48 [97.0 to 99.9]
  G12: 35 minutes | 99.69 [96.2 to 100.0]

13. Primary Outcome: Part 2, Group 3, Cohort 2J: Median Percentage of Gluten Degradation by PvP001 900 mg in a Standardized 6 gm Gluten-containing Study Meal at 65 Minutes After Administration of PvP001
Description: as for outcome 6
Time Frame: Cohort Treatment Day: at 65 minutes post-dose
Population: as for outcome 11
Measure: Median (Full Range); unit: percentage of gluten degradation
Arm/Group | Part 2, Group 3: PvP001 900 mg (2J)
Number analyzed (Participants) | 8
percentage of gluten degradation
  R5: 65 minutes | 99.22 [87.8 to 100.0]
  G12: 65 minutes | 98.49 [76.1 to 100.0]

14. Primary Outcome: Part 3, Groups 1 to 5, Cohorts 3B, 3D, 3F, 3H and 3J: Median Percentage of Gluten Degradation by PvP003 150 mg and 600 mg in a Standardized 1 gm Gluten-containing Study Meal at 35 Minutes After Administration of PvP003
Description: as for outcome 6
Time Frame: Cohort Treatment Day: at 35 minutes
Population: ITT population in Part 3 of study, included all participants who received at least one dose of study drug. As planned, this outcome measure was assessed for Group 1, Cohort 3B (PvP003 600 mg), Group 2, Cohort 3D (PvP003 600 mg), Group 3, Cohort 3F (PvP003 600 mg), Group 4, Cohort 3H (PvP003 600 mg) and Group 5, Cohort 3J (PvP003 150 mg) of Part 3. Here 'N' (overall number of participants analyzed) included all participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: percentage of gluten degradation
Groups:
- Part 3, Group 1: PvP003 600 mg (3B): PvP003 (TAK-062 tablet formulation) 600 mg (3B) with pretreatment buffer solution administered prior to the PvP003 before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3B in healthy participants.
- Part 3, Group 2: PvP003 600 mg (3D): PvP003 (TAK-062 tablet formulation) 600 mg (3D) without pretreatment buffer solution before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3D in healthy participants.
- Part 3, Group 3: PvP003 600 mg (3F): PvP003 (TAK-062 tablet formulation) 600 mg (3F) without pretreatment buffer solution administered after an approximately 50 mL portion of standardized 1 gram gluten-containing study meal and then remaining portion of the 1 gram gluten-containing study meal was ingested after administration of PvP0003, orally, single dose on Cohort Treatment Day of Cohort 3F in healthy participants.
- Part 3, Group 4: PvP003 600 mg (3H): PvP003 (TAK-062 tablet formulation) 600 mg (3H) without pretreatment buffer solution before standardized gluten-free study meal followed by a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3H in healthy participants.
- Part 3, Group 5: PvP003 150 mg (3J): PvP003 (TAK-062 tablet formulation) 150 mg (3J) without pretreatment buffer solution before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3J in healthy participants.
Arm/Group | Part 3, Group 1: PvP003 600 mg (3B) | Part 3, Group 2: PvP003 600 mg (3D) | Part 3, Group 3: PvP003 600 mg (3F) | Part 3, Group 4: PvP003 600 mg (3H) | Part 3, Group 5: PvP003 150 mg (3J)
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 12
percentage of gluten degradation
  R5: 35 minutes | 94.68 [57.0 to 97.5] | 79.69 [-17.0 to 95.4] | 68.49 [26.6 to 98.9] | NA [NA to NA] — Data was not estimable due to gluten concentrations below the limit of quantification (LLOQ) of 10 microgram per milliliter (mcg/mL). | 88.23 [-970.5 to 99.7]
  G12: 35 minutes | 96.66 [73.5 to 99.2] | 71.71 [-24.5 to 96.5] | 71.11 [-200.0 to 96.0] | NA [NA to NA] — Data was not estimable due to gluten concentrations below the limit of quantification (LLOQ) of 10 microgram per milliliter (mcg/mL). | 93.12 [-554.2 to 99.7]

15. Primary Outcome: Part 3, Groups 1 to 5, Cohorts 3B, 3D, 3F, 3H and 3J: Median Percentage of Gluten Degradation by PvP003 150 mg and 600 mg in a Standardized 1 gm Gluten-containing Study Meal at 65 Minutes After Administration of PvP003
Description: as for outcome 6
Time Frame: Cohort Treatment Day: at 65 minutes
Population: ITT population in Part 3 of study, included all participants who received at least one dose of study drug. As planned, this outcome measure was assessed for Group 1, Cohort 3B (PvP003 600 mg), Group 2, Cohort 3D (PvP003 600 mg), Group 3, Cohort 3F (PvP003 600 mg), Group 4,Cohort 3H (PvP003 600 mg), Group 5, Cohort 3J (PvP003 150 mg) of Part 3. Here 'N' (overall number of participants analyzed) included all participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: percentage of gluten degradation
Arm/Group | Part 3, Group 1: PvP003 600 mg (3B) | Part 3, Group 2: PvP003 600 mg (3D) | Part 3, Group 3: PvP003 600 mg (3F) | Part 3, Group 4: PvP003 600 mg (3H) | Part 3, Group 5: PvP003 150 mg (3J)
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 12
percentage of gluten degradation
  R5: 65 minutes | 89.54 [-1082.4 to 99.8] | 50.36 [-149.1 to 95.1] | 85.63 [47.4 to 99.1] | 98.86 [-252.0 to 99.8] | 84.48 [-312.3 to 99.8]
  G12: 65 minutes | 95.34 [-899.5 to 99.6] | 64.40 [-91.2 to 96.6] | 85.69 [-39.5 to 98.7] | 96.34 [-224.1 to 98.6] | 92.35 [-423.2 to 99.8]

16. Secondary Outcome: Part 1 and Part 2, Cmax: Maximum Observed Plasma Concentration for PvP001 and PvP002
Time Frame: Cohort Treatment Day pre-dose and at multiple time points (up to 480 minutes) post-dose
Population: Pharmacokinetic (PK) population included all participants who received at least one dose of study drug and had any PK data. As planned, this outcome measure was to be assessed for Parts 1 and 2 PvP001 and PvP002; however, PK analysis was not conducted since plasma concentrations were below the LLOQ at all sampling time-points for all arms.
Groups:
- Part 1, (1E-1): PvP002 600 mg: PvP001 (TAK-062 capsule formulation) 600 mg, orally, single dose on Cohort Treatment Day in healthy participants.
- Part 1, (1E-2): PvP002 600 mg: PvP001 (TAK-062 capsule formulation) 600 mg, orally, single dose on Cohort Treatment Day in CeD participants.
- Part 2, Group 2: PvP002 Placebo (2D): PvP002 comparator (sterile water) (2D), orally, single dose on Cohort Treatment Day of Cohort 2D in healthy participants.
Arm/Group | Part 1, (1B-1): PvP001 100 mg | Part 1, (1C-1): PvP001 300 mg | Part 1, (1D-1): PvP001 900 mg | Part 1, (1E-1): PvP002 600 mg | Part 1, (1B-2): PvP001 100 mg | Part 1, (1C-2): PvP001 300 mg | Part 1, (1D-2): PvP001 900 mg | Part 1, (1E-2): PvP002 600 mg | Part 2, Group 1: PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg With PPI (2C) | Part 2, Group 2: PvP002 Placebo (2D) | Part 2, Group 2: PvP002 600 mg (2E) | Part 2, Group 3: PvP001 300 mg (2G) | Part 2, Group 3: PvP001 600 mg (2H) | Part 2, Group 3: PvP001 900 mg (2J)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Part 1 and Part 2, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for PvP001 and PvP002
Time Frame: Cohort Treatment Day pre-dose and at multiple time points (up to 480 minutes) post-dose
Population: PK population included all participants who received at least one dose of study drug and had any PK data. As planned, this outcome measure was to be assessed for Parts 1 and 2 PvP001 and PvP002; however, PK analysis was not conducted since plasma concentrations were below the LLOQ at all sampling time-points for all arms.
Arm/Group | Part 1, (1B-1): PvP001 100 mg | Part 1, (1C-1): PvP001 300 mg | Part 1, (1D-1): PvP001 900 mg | Part 1, (1E-1): PvP002 600 mg | Part 1, (1B-2): PvP001 100 mg | Part 1, (1C-2): PvP001 300 mg | Part 1, (1D-2): PvP001 900 mg | Part 1, (1E-2): PvP002 600 mg | Part 2, Group 1: PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg With PPI (2C) | Part 2, Group 2: PvP002 Placebo (2D) | Part 2, Group 2: PvP002 600 mg (2E) | Part 2, Group 3: PvP001 300 mg (2G) | Part 2, Group 3: PvP001 600 mg (2H) | Part 2, Group 3: PvP001 900 mg (2J)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Part 1 and Part 2, T(1/2): Terminal Disposition Phase Half-life of PvP001 and PvP002
Time Frame: Cohort Treatment Day pre-dose and at multiple time points (up to 480 minutes) post-dose
Population: as for outcome 17
Arm/Group | Part 1, (1B-1): PvP001 100 mg | Part 1, (1C-1): PvP001 300 mg | Part 1, (1D-1): PvP001 900 mg | Part 1, (1E-1): PvP002 600 mg | Part 1, (1B-2): PvP001 100 mg | Part 1, (1C-2): PvP001 300 mg | Part 1, (1D-2): PvP001 900 mg | Part 1, (1E-2): PvP002 600 mg | Part 2, Group 1: PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg With PPI (2C) | Part 2, Group 2: PvP002 Placebo (2D) | Part 2, Group 2: PvP002 600 mg (2E) | Part 2, Group 3: PvP001 300 mg (2G) | Part 2, Group 3: PvP001 600 mg (2H) | Part 2, Group 3: PvP001 900 mg (2J)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Part 1 and Part 2, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for PvP001 and PvP002
Time Frame: Cohort Treatment Day pre-dose and at multiple time points (up to 480 minutes) post-dose
Population: as for outcome 17
Arm/Group | Part 1, (1B-1): PvP001 100 mg | Part 1, (1C-1): PvP001 300 mg | Part 1, (1D-1): PvP001 900 mg | Part 1, (1E-1): PvP002 600 mg | Part 1, (1B-2): PvP001 100 mg | Part 1, (1C-2): PvP001 300 mg | Part 1, (1D-2): PvP001 900 mg | Part 1, (1E-2): PvP002 600 mg | Part 2, Group 1: PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg With PPI (2C) | Part 2, Group 2: PvP002 Placebo (2D) | Part 2, Group 2: PvP002 600 mg (2E) | Part 2, Group 3: PvP001 300 mg (2G) | Part 2, Group 3: PvP001 600 mg (2H) | Part 2, Group 3: PvP001 900 mg (2J)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Part 1 and Part 2, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for PvP001 and PvP002
Time Frame: Cohort Treatment Day pre-dose and at multiple time points (up to 480 minutes) post-dose
Population: as for outcome 17
Arm/Group | Part 1, (1B-1): PvP001 100 mg | Part 1, (1C-1): PvP001 300 mg | Part 1, (1D-1): PvP001 900 mg | Part 1, (1E-1): PvP002 600 mg | Part 1, (1B-2): PvP001 100 mg | Part 1, (1C-2): PvP001 300 mg | Part 1, (1D-2): PvP001 900 mg | Part 1, (1E-2): PvP002 600 mg | Part 2, Group 1: PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg With PPI (2C) | Part 2, Group 2: PvP002 Placebo (2D) | Part 2, Group 2: PvP002 600 mg (2E) | Part 2, Group 3: PvP001 300 mg (2G) | Part 2, Group 3: PvP001 600 mg (2H) | Part 2, Group 3: PvP001 900 mg (2J)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Part 1 and Part 2: Number of Participants With Anti-drug Antibodies (ADA) for PvP001 and PvP002
Time Frame: At Day 14 and Day 28
Population: Safety population included all participants who received at least one dose of study drug. As planned, data was collected and analyzed at Day 14 and Day 28 after the final Cohort Treatment Day to test for ADA to PvP001 and PvP002; therefore, sequence-wise data is reported for Parts 1 and 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, (1A-1): PvP001 Placebo | Part 1, (1B-1): PvP001 100 mg | Part 1, (1C-1): PvP001 300 mg | Part 1, (1D-1): PvP001 900 mg | Part 1, (1E-1): PvP002 600 mg | Part 1, (1A-2): PvP001 Placebo | Part 1, (1B-2): PvP001 100 mg | Part 1, (1C-2): PvP001 300 mg | Part 1, (1D-2): PvP001 900 mg | Part 1, (1E-2): PvP002 600 mg | Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) | Part 2, Group 1: PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg (2B) + PvP001 Placebo (2A) + PvP001 900 mg With PPI (2C) | Part 2, Group 1: PvP001 900 mg (2B) + PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) | Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 Placebo (2A) + PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg With PPI (2C) + PvP001 900 mg (2B) + PvP001 Placebo (2A) | Part 2, Group 2: PvP002 Comparator (2D) + PvP002 600 mg (2E) | Part 2, Group 2: PvP002 600 mg (2E) + PvP002 Comparator (2D) | Part 2, Group 3: PvP001 Placebo (2F) + PvP001 300 mg (2G) | Part 2, Group 3: PvP001 300 mg (2G) + PvP001 Placebo (2F) | Part 2, Group 3: PvP001 Placebo (2F) + PvP001 600 mg (2H) | Part 2, Group 3: PvP001 600 mg (2H) + PvP001 Placebo (2F) | Part 2, Group 3: PvP001 Placebo (2I) + PvP001 900 mg (2J) | Part 2, Group 3: PvP001 900 mg (2J) + PvP001 Placebo (2I)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 1 | 3 | 3 | 2 | 2 | 2 | 2 | 4 | 5 | 4 | 4 | 4 | 4 | 4 | 4
Participants
  Day 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Part 1: Maximum Tolerated Dose (MTD) of PvP001
Description: MTD was defined as the maximum dose that was determined to be safe and tolerable for Part 1 (1B-1 and 1B-2, 1C-1 and 1C-2, 1D-1 and 1D-2) in healthy or CeD participants.
Time Frame: Cohort Treatment Day up to Day 7
Population: Safety population included all participants who received at least one dose of study drug. As planned, this outcome measure was assessed only for Part 1 (1B-1 and 1B-2, 1C-1 and 1C-2, 1D-1 and 1D-2) in healthy or CeD participants of the study. Here 'N' (overall number of participants analyzed) included all participants who were evaluable for this outcome measure.
Measure: Number; unit: mg
Groups:
- Part 1: PVP001 (TAK-062 Liquid Formulation) All Cohorts: PVP001 (TAK-062 liquid formulation) 100mg for 1B-1 and 1B-2, 300 mg for 1C-1 and 1C-2, 900 mg for 1D-1 and 1D-2, orally, single dose on Cohort Treatment Day of each cohort in healthy or CeD participants.
Arm/Group | Part 1: PVP001 (TAK-062 Liquid Formulation) All Cohorts
Number analyzed (Participants) | 22
mg | 900

23. Secondary Outcome: Part 2: Number of Participants Reporting One or More TEAEs and TESAEs for PvP001 and PvP002
Time Frame: Cohort Treatment Day up to 5 days after the final Cohort Treatment Day (up to Day 22)
Population: Safety population included all participants who received at least one dose of study drug. As planned, this outcome measure was assessed only in the Part 2 of this study.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2, Group 1: PvP001 Placebo (2A): PvP001 (TAK-062 liquid formulation) placebo-matching liquid (2A), orally, single dose on Cohort Treatment Day of Cohort 2A in healthy participants.
- Part 2, Group 2: PvP002 Comparator (2D): PvP002 capsule comparator (sterile water) (2D), orally, single dose on Cohort Treatment Day of Cohort 2D in healthy participants.
- Part 2, Group 3: PvP001 Placebo (2F and 2I): PvP001 (TAK-062 liquid formulation) placebo-matching liquid (2F), orally, single dose on Cohort Treatment Day of Cohort 2F and 2I in healthy participants.
Arm/Group | Part 2, Group 1: PvP001 Placebo (2A) | Part 2, Group 1: PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg With PPI (2C) | Part 2, Group 2: PvP002 Comparator (2D) | Part 2, Group 2: PvP002 600 mg (2E) | Part 2, Group 3: PvP001 Placebo (2F and 2I) | Part 2, Group 3: PvP001 300 mg (2G) | Part 2, Group 3: PvP001 600 mg (2H) | Part 2, Group 3: PvP001 900 mg (2J)
Number analyzed (Participants) | 13 | 12 | 13 | 9 | 9 | 24 | 8 | 8 | 8
Participants
  TEAEs | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0
  TESAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Part 3: Number of Participants Reporting One or More TEAEs and TESAEs With PvP003 After a Single Dose
Time Frame: Cohort Treatment Day up to 5 days after final Cohort Treatment Day (up to Day 10)
Population: Safety population included all participants who received at least one dose of study drug. As planned, this outcome measure was assessed for Part 3 of this study.
Measure: Count of Participants; unit: Participants
Groups:
- Part 3, Group 1: PvP003 Placebo (3A, 3C, 3E, 3G and 3I): PvP003 (TAK-062 tablet formulation) placebo-matching tablet orally, single dose on Cohorts Treatment Day of 3A, 3C, 3E, 3G or 3I in healthy participants. For Cohort 3A: with pretreatment buffer solution administered prior to the PvP003 before a standardized 1 gm gluten-containing study meal. For Cohorts 3C and 3I: without pretreatment buffer solution before a standardized 1 gm gluten-containing study meal. For Cohort 3E: without pretreatment buffer solution administered after an approximately 50 mL portion of standardized 1 gram gluten-containing study meal and then remaining portion of the 1 gram gluten-containing study meal was ingested after administration of PvP0003; and for Cohort 3G: without pretreatment buffer solution before standardized gluten-free study meal followed by a standardized 1 gm gluten-containing study meal.
Arm/Group | Part 3, Group 1: PvP003 Placebo (3A, 3C, 3E, 3G and 3I) | Part 3, Group 1: PvP003 600 mg (3B) | Part 3, Group 2: PvP003 600 mg (3D) | Part 3, Group 3: PvP003 600 mg (3F) | Part 3, Group 4: PvP003 600 mg (3H) | Part 3, Group 5: PvP003 150 mg (3J)
Number analyzed (Participants) | 36 | 6 | 6 | 6 | 6 | 13
Participants
  TEAEs | 4 | 1 | 0 | 0 | 1 | 1
  TESAEs | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Part 3, Cmax: Maximum Observed Plasma Concentration for PvP003 150 mg and 600 mg Single Dose
Time Frame: Cohort Treatment Day pre-dose and at multiple time points (up to 480 minutes) post-dose
Population: PK population included all participants who received at least one dose of study drug and had any PK data. As planned, this outcome measure was to be assessed for Part 3, PvP003 150 mg and 600 mg cohorts; however, PK analysis was not conducted since plasma concentrations were below the LLOQ at all sampling time-points for all arms.
Groups:
- Part 3, Group 1: PvP003 600 mg (3B): PvP003 (TAK-062 tablet formulation) 600 mg (3B) with pretreatment buffer solution with pretreatment buffer solution administered prior to the PvP003 before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3B in healthy participants.
Arm/Group | Part 3, Group 1: PvP003 600 mg (3B) | Part 3, Group 2: PvP003 600 mg (3D) | Part 3, Group 3: PvP003 600 mg (3F) | Part 3, Group 4: PvP003 600 mg (3H) | Part 3, Group 5: PvP003 150 mg (3J)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Part 3, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for PvP003 150 mg and 600 mg Single Dose
Time Frame: Cohort Treatment Day pre-dose and at multiple time points (up to 480 minutes) post dose
Population: as for outcome 25
Groups:
- Part 3, Group 3: PvP003 600 mg (3F): PvP003 (TAK-062 tablet formulation) 600 mg (3F) without pretreatment buffer solution administered after an approximately 50 mL portion of standardized 1 gram gluten-containing study meal and then remaining portion of the 1 gram gluten-containing study meal was ingested after administration of PvP0003, single dose on Cohort Treatment Day of Cohort 3F in healthy participants.
Arm/Group | Part 3, Group 1: PvP003 600 mg (3B) | Part 3, Group 2: PvP003 600 mg (3D) | Part 3, Group 3: PvP003 600 mg (3F) | Part 3, Group 4: PvP003 600 mg (3H) | Part 3, Group 5: PvP003 150 mg (3J)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Part 3, T(1/2): Terminal Disposition Phase Half-life of PvP003 150 mg and 600 mg Single Dose
Time Frame: Cohort Treatment Day pre-dose and at multiple time points (up to 480 minutes) post dose
Population: as for outcome 25
Arm/Group | Part 3, Group 1: PvP003 600 mg (3B) | Part 3, Group 2: PvP003 600 mg (3D) | Part 3, Group 3: PvP003 600 mg (3F) | Part 3, Group 4: PvP003 600 mg (3H) | Part 3, Group 5: PvP003 150 mg (3J)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Part 3, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for PvP003 150 mg and 600 mg Single Dose
Time Frame: Cohort Treatment Day pre-dose and at multiple time points (up to 480 minutes) post dose
Population: as for outcome 25
Arm/Group | Part 3, Group 1: PvP003 600 mg (3B) | Part 3, Group 2: PvP003 600 mg (3D) | Part 3, Group 3: PvP003 600 mg (3F) | Part 3, Group 4: PvP003 600 mg (3H) | Part 3, Group 5: PvP003 150 mg (3J)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

29. Secondary Outcome: Part 3, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for PvP003 150 mg and 600 mg Single Dose
Time Frame: Cohort Treatment Day pre-dose and at multiple time points (up to 480 minutes) post dose
Population: as for outcome 25
Arm/Group | Part 3, Group 1: PvP003 600 mg (3B) | Part 3, Group 2: PvP003 600 mg (3D) | Part 3, Group 3: PvP003 600 mg (3F) | Part 3, Group 4: PvP003 600 mg (3H) | Part 3, Group 5: PvP003 150 mg (3J)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Part 3: Number of Participants With ADA for PvP003 150 mg and 600 mg Single Dose
Time Frame: At Day 14 and Day 28
Population: Safety population included all participants who received at least one dose of study drug. As planned, this outcome measure was assessed only for Part 3 of this study. As planned, data was collected and analyzed at Day 14 and Day 28 after the final Cohort Treatment Day to test for ADA to PvP003; therefore, sequence-wise data is reported for Part 3.
Measure: Count of Participants; unit: Participants
Groups:
- Part 3, Group 3: PvP003 Placebo (3E) + PvP003 600 mg (3F): PvP003 (TAK-062 tablet formulation) placebo-matching tablet (3E) without pretreatment buffer solution administered after an approximately 50 mL portion of standardized 1 gram gluten-containing study meal and then remaining portion of the 1 gram gluten-containing study meal was ingested after administration of PvP0003, orally, single dose on Cohort Treatment Day of Cohort 3E, followed by PvP003 600 mg (3F) without pretreatment buffer solution administered after an approximately 50 mL portion of standardized 1 gram gluten-containing study meal and then remaining portion of the 1 gram gluten-containing study meal was ingested after administration of PvP0003, orally, single dose on Cohort Treatment Day of Cohort 3F in healthy participants. There was a washout period of 3 days between each Cohort Treatment Day.
- Part 3, Group 3: PvP003 600 mg (3F) + PvP003 Placebo (3E): PvP003 (TAK-062 tablet formulation) 600 mg (3F) without pretreatment buffer solution before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3F, followed by PvP003 placebo-matching tablet (3E) without pretreatment buffer solution before a standardized 1 gm gluten-containing study meal, orally, single dose on Cohort Treatment Day of Cohort 3E, in healthy participants. There was a washout period of 3 days between each Cohort Treatment Day.
Arm/Group | Part 3, Group 1: PvP003 Placebo (3A) + PvP003 600 mg (3B) | Part 3, Group 1: PvP003 600 mg (3B) + PvP003 Placebo (3A) | Part 3, Group 2: PvP003 Placebo (3C) + PvP003 600 mg (3D) | Part 3, Group 2: PvP003 600 mg (3D) + PvP003 Placebo (3C) | Part 3, Group 3: PvP003 Placebo (3E) + PvP003 600 mg (3F) | Part 3, Group 3: PvP003 600 mg (3F) + PvP003 Placebo (3E) | Part 3, Group 4: PvP003 Placebo (3G) + PvP003 600 mg (3H) | Part 3, Group 4: PvP003 600 mg (3H) + PvP003 Placebo (3G) | Part 3, Group 5: PvP003 Placebo (3I) + PvP003 150 mg (3J) | Part 3, Group 5: PvP003 150 mg (3J) + PvP003 Placebo (3I)
Number analyzed (Participants) | 3 | 4 | 1 | 5 | 3 | 3 | 3 | 3 | 5 | 8
Participants
  Day 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

31. Secondary Outcome: Part 4, Cmax: Maximum Observed Plasma Concentration for PvP003 600 mg Multiple Dose
Time Frame: Cohort Treatment Days 1 and 5 pre-dose and at multiple time points (up to 240 minutes) post dose
Population: PK population included all participants who received at least one dose of study drug and had any PK data. As planned, this outcome measure was to be assessed for Part 4, PvP003 600 mg, TID (4B); however, PK analysis was not conducted since plasma concentrations were below the LLOQ at all sampling time-points for all arms.
Arm/Group | Part 4: PvP003 600 mg, TID (4B)
Number analyzed (Participants) | 0

32. Secondary Outcome: Part 4, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for PvP003 600 mg Multiple Dose
Time Frame: Cohort Treatment Days 1 and 5 pre-dose and at multiple time points (up to 240 minutes) post dose
Population: PK population included all participants who received at least one dose of study drug and had any PK data. As planned, this outcome measure was to be assessed for Part 4, PvP003 600 mg, TID (4B); however, PK analysis was not conducted since plasma concentrations were below the LLOQ at all sampling time points for all arms.
Arm/Group | Part 4: PvP003 600 mg, TID (4B)
Number analyzed (Participants) | 0

33. Secondary Outcome: Part 4, T(1/2): Terminal Disposition Phase Half-life of PvP003 600 mg Multiple Dose
Time Frame: Cohort Treatment Days 1 and 5 pre-dose and at multiple time points (up to 240 minutes) post dose
Population: as for outcome 32
Arm/Group | Part 4: PvP003 600 mg, TID (4B)
Number analyzed (Participants) | 0

34. Secondary Outcome: Part 4, AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for PvP003 600 mg Multiple Dose
Time Frame: Cohort Treatment Days 1 and 5 pre-dose and at multiple time points (up to 240 minutes) post dose
Population: as for outcome 32
Arm/Group | Part 4: PvP003 600 mg, TID (4B)
Number analyzed (Participants) | 0

35. Secondary Outcome: Part 4, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for PvP003 600 mg Multiple Dose
Time Frame: Cohort Treatment Days 1 and 5 pre-dose and at multiple time points (up to 240 minutes) post dose
Population: as for outcome 32
Arm/Group | Part 4: PvP003 600 mg, TID (4B)
Number analyzed (Participants) | 0

36. Secondary Outcome: Part 4: Number of Participants With ADA for PvP003 600 mg Multiple Dose
Time Frame: At Day 14 and Day 28
Population: Safety population included all participants who received at least one dose of study drug. As planned, this outcome measure was assessed only for Part 4 of this study. As planned, data was collected and analyzed at Day 14 and Day 28 after Day 5 of the second Cohort Treatment Period to test for ADA to PvP003; therefore, sequence-wise data is reported for Part 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 4: PvP003 Placebo, TID (4A) + PvP003 600 mg, TID (4B) | Part 4: PvP003 600 mg, TID (4B) + PvP003 Placebo, TID (4A)
Number analyzed (Participants) | 3 | 3
Participants
  Day 14 | 1 | 1
  Day 28 | 1 | 0

ADVERSE EVENTS:
Time Frame: TEAEs were adverse events that started after the first dose of study drug in Part 1, 2, 3 and 4: Cohort Treatment Day up to 5 days after 24-hour safety assessment on Day 2 (up to Day 7) in Part 1; Cohort Treatment Day up to 5 days after the final Cohort Treatment Day (up to Day 22 in Part 2, and up to Day 10 in Part 3); and Day 1 of Cohort Treatment Period 1 up to 5 days after the Day 5 of Cohort Treatment Period 2 (up Day 28) in Part 4
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Part 3, Group 1: PvP003 Placebo (3A, 3C, 3E, 3G and 3I): PvP003 (TAK-062 tablet formulation) placebo-matching tablet orally, single dose on Cohorts Treatment Day 1 of 3A, 3C, 3E, 3G or 3I in healthy participants. For Cohort 3A: with pretreatment buffer solution administered prior to the PvP003 before a standardized 1 gm gluten-containing study meal. For Cohorts 3C and 3I: without pretreatment buffer solution before a standardized 1 gm gluten-containing study meal. For Cohort 3E: without pretreatment buffer solution administered after an approximately 50 mL portion of standardized 1 gram gluten-containing study meal and then remaining portion of the 1 gram gluten-containing study meal was ingested after administration of PvP0003; and for Cohort 3G: without pretreatment buffer solution before standardized gluten-free study meal followed by a standardized 1 gm gluten-containing study meal.
Arm/Group | Part 1, (1A-1): PvP001 Placebo | Part 1, (1B-1): PvP001 100 mg | Part 1, (1C-1): PvP001 300 mg | Part 1, (1D-1): PvP001 900 mg | Part 1, (1E-1): PvP002 600 mg | Part 1, (1A-2): PvP001 Placebo | Part 1, (1B-2): PvP001 100 mg | Part 1, (1C-2): PvP001 300 mg | Part 1, (1D-2): PvP001 900 mg | Part 1, (1E-2): PvP002 600 mg | Part 2, Group 1: PvP001 Placebo (2A) | Part 2, Group 1: PvP001 900 mg (2B) | Part 2, Group 1: PvP001 900 mg With PPI (2C) | Part 2, Group 2: PvP002 Comparator (2D) | Part 2, Group 2: PvP002 600 mg (2E) | Part 2, Group 3: PvP001 Placebo (2F and 2I) | Part 2, Group 3: PvP001 300 mg (2G) | Part 2, Group 3: PvP001 600 mg (2H) | Part 2, Group 3: PvP001 900 mg (2J) | Part 3, Group 1: PvP003 Placebo (3A, 3C, 3E, 3G and 3I) | Part 3, Group 1: PvP003 600 mg (3B) | Part 3, Group 2: PvP003 600 mg (3D) | Part 3, Group 3: PvP003 600 mg (3F) | Part 3, Group 4: PvP003 600 mg (3H) | Part 3, Group 5: PvP003 150 mg (3J) | Part 4: PvP003 Placebo, TID (4A) | Part 4: PvP003 600 mg, TID (4B)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/1 | 0/13 | 0/12 | 0/13 | 0/9 | 0/9 | 0/24 | 0/8 | 0/8 | 0/8 | 0/36 | 0/6 | 0/6 | 0/6 | 0/6 | 0/13 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/1 | 0/13 | 0/12 | 0/13 | 0/9 | 0/9 | 0/24 | 0/8 | 0/8 | 0/8 | 0/35 | 0/6 | 0/6 | 0/6 | 0/6 | 0/13 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 3/3 | 0/3 | 2/3 | 1/3 | 1/1 | 1/13 | 0/12 | 2/13 | 0/9 | 0/9 | 1/24 | 1/8 | 1/8 | 0/8 | 4/36 | 1/6 | 0/6 | 0/6 | 1/6 | 1/13 | 0/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, (1A-1): PvP001 Placebo (N=3) | Part 1, (1B-1): PvP001 100 mg (N=3) | Part 1, (1C-1): PvP001 300 mg (N=3) | Part 1, (1D-1): PvP001 900 mg (N=3) | Part 1, (1E-1): PvP002 600 mg (N=3) | Part 1, (1A-2): PvP001 Placebo (N=3) | Part 1, (1B-2): PvP001 100 mg (N=3) | Part 1, (1C-2): PvP001 300 mg (N=3) | Part 1, (1D-2): PvP001 900 mg (N=3) | Part 1, (1E-2): PvP002 600 mg (N=1) | Part 2, Group 1: PvP001 Placebo (2A) (N=13) | Part 2, Group 1: PvP001 900 mg (2B) (N=12) | Part 2, Group 1: PvP001 900 mg With PPI (2C) (N=13) | Part 2, Group 2: PvP002 Comparator (2D) (N=9) | Part 2, Group 2: PvP002 600 mg (2E) (N=9) | Part 2, Group 3: PvP001 Placebo (2F and 2I) (N=24) | Part 2, Group 3: PvP001 300 mg (2G) (N=8) | Part 2, Group 3: PvP001 600 mg (2H) (N=8) | Part 2, Group 3: PvP001 900 mg (2J) (N=8) | Part 3, Group 1: PvP003 Placebo (3A, 3C, 3E, 3G and 3I) (N=36) | Part 3, Group 1: PvP003 600 mg (3B) (N=6) | Part 3, Group 2: PvP003 600 mg (3D) (N=6) | Part 3, Group 3: PvP003 600 mg (3F) (N=6) | Part 3, Group 4: PvP003 600 mg (3H) (N=6) | Part 3, Group 5: PvP003 150 mg (3J) (N=13) | Part 4: PvP003 Placebo, TID (4A) (N=6) | Part 4: PvP003 600 mg, TID (4B) (N=6)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT03701555/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT03701555/SAP_001.pdf